CLINICAL TRIAL: NCT03561519
Title: FECAL MICROBIOTA TRANSPLANTATION IN THE TREATMENT OF IRRITABLE BOWEL SYNDROME
Brief Title: FMT in the Treatment of IBS
Acronym: FMT-IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joint Authority for Päijät-Häme Social and Health Care (Other)
Collaborators: Helsinki University Central Hospital (Other); University of Helsinki (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 40/13/03/01/15
Record Dates: First submitted 2018-06-06; First posted 2018-06-19 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-06

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Placebo controlled trial. 50% of patients received autologous FMT as placebo and 50% received FMT from a healthy donor.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization was done by personnel not treating the patient. The participant or FMT providing personnel did not know the result of randomization. The doctors assessing the outcome have been blinded of the result of randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT (Active Comparator): IBS patients randomized to receive FMT from a healthy donor.
  Interventions: Other: Fecal Microbiota Transplantation (FMT)
- Placebo (Placebo Comparator): IBS patients randomized to receive autologous FMT (fecal suspension made of their own feces) as a placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Fecal Microbiota Transplantation (FMT) — Fecal suspension administered in colonoscopy into the cecum of the patient.
  Arms: FMT
Other: Placebo — As a placebo a fecal suspension made of patients own feces is administered into the cecum of the patient in colonoscopy.
  Arms: Placebo

SUMMARY:
52 adult IBS patients were recruited. 50% were given a fecal microbiota transplantation in colonoscopy and 50% were given an FMT made of their own feces as placebo. follow up time was 1 year after FMT.

DETAILED DESCRIPTION:
52 adult IBS patients of any subgroup(IBS-D, IBS-C or IBS-M), were recruited and given an FMT in colonoscopy. Neither the patient nor the care taking personnel did know in which group the patients belonged to. The patients were screened with fecal samples for 16RNA sequencing and they were repeatedly done IBS-SSS questionnaire and questionnaires for quality of life and psychical condition. Follow up time was 1 year after the colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IBS based on Rome III criteria
* Having received traditional treatment for at least 1 month
* Availability of consecutive fecal samples over one year.
* Compliance to attend ileocolonoscopy and FMT procedure.
* 18-75 years

Exclusion Criteria:

* Unable to provide informed consent
* Antibiotic therapy in past 3 months
* Inflammatory bowel disease (IBD)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-08-27 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
IBS symptom relieve | 52 weeks
  Reduction IBS-SSS by 50 points, The irritable bowel severity score system in which the maximum achievable score is 500. Mild, moderate and severe cases are indicated by scores of 75 to 175, 175 to 300 and > 300.( Aliment Pharmacol Ther. 1997 Apr;11(2):395-402.)

CONTACTS AND LOCATIONS:
Overall Officials: Perttu Arkkila, Adj. Prof., Study Chair — +358 9 4711
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- [Derived] Lahtinen P, Jalanka J, Hartikainen A, Mattila E, Hillila M, Punkkinen J, Koskenpato J, Anttila VJ, Tillonen J, Satokari R, Arkkila P. Randomised clinical trial: faecal microbiota transplantation versus autologous placebo administered via colonoscopy in irritable bowel syndrome. Aliment Pharmacol Ther. 2020 Jun;51(12):1321-1331. doi: 10.1111/apt.15740. Epub 2020 Apr 28. PMID 32343000